CLINICAL TRIAL: NCT03404310
Title: Oral Zinc Sulfate for the Treatment of High Risk Cervical HPV Versus Placebo
Brief Title: Zinc Sulfate for Human Papillomavirus (HPV)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPV-Zinc
Record Dates: First submitted 2017-11-27; First posted 2018-01-19 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Human Papilloma Virus
Keywords: HPV; ASCUS; LSIL; Cervical Cancer
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix; Uterine Cervical Neoplasms | interventions — Zinc Sulfate; Gelatin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded placebo controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Zinc Sulfate 220mg twice daily for three months.
  Interventions: Dietary Supplement: Zinc Sulfate
- Placebo (Placebo Comparator): Gelatin Placebo tablet twice daily for three months.
  Interventions: Other: Placebo (Gelatin Tablet)

INTERVENTIONS:
Dietary Supplement: Zinc Sulfate — Participant will take one 220mg tablet twice daily for three months.
  Arms: Treatment
Other: Placebo (Gelatin Tablet) — Participant will take one tablet twice daily for three months.
  Arms: Placebo

SUMMARY:
The Human Papillomavirus (HPV) is well established as the primary causative agent in both warts and cervical cancer. Although cervical high risk HPV (hrHPV) infections have a high rate of spontaneous resolution this takes time and the infection can cause cervical cells to progress to precancerous and cancerous lesions. Zinc has been shown to play a central role in immunity. This study is to determine if oral zinc sulfate can improve clearance rates of high risk HPV versus placebo.

DETAILED DESCRIPTION:
Upon enrollment eligible participants will be randomized and given a three-month supply of zinc sulfate or placebo to be taken as directed. They will have zinc serum lab testing at enrollment and upon study completion. Patients will also be asked to complete short questionnaires and to make study staff aware of any side effects they should experience.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal cytology of atypical squamous cells of undetermined significance (ASCUS) on Pap smear OR
* Low-grade squamous intra epithelial lesions (LSIL) on Pap smear OR
* Positive hrHPV on routine screening (positive HPV will be assumed to be high grade)

Exclusion Criteria:

* Patients who proceed to excisional procedures (loop electrosurgical excision procedure or cold knife conization)
* Pregnant patients
* Breastfeeding patients
* Immunocompromised patients

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Clearance rates of high risk HPV | During 3 month treatment period

SECONDARY OUTCOMES:
Progression versus Regression | During 3 month treatment period
  Incidence of progression versus regression of cervical changes after treatment with oral zinc sulfate
Side Effects | After 3 month treatment period
  Rates of side effects from zinc sulfate
Compliance Rates | After 3 month treatment period
  Examine rates of patients finishing the 3-month course of zinc sulfate
Parity | After 3 month treatment period
  Examine the correlation of parity on HPV clearance
Low Zinc Levels and Persistence | After 3 month treatment period
  Examine potential correlation between low serum levels of zinc and persistence of HPV.
Zinc Levels and Regression | After 3 month treatment period
  Examine the relation between zinc levels before and after treatment and the relation to regression of HPV.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Prudnick, DO, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Sanjose S, Quint WG, Alemany L, Geraets DT, Klaustermeier JE, Lloveras B, Tous S, Felix A, Bravo LE, Shin HR, Vallejos CS, de Ruiz PA, Lima MA, Guimera N, Clavero O, Alejo M, Llombart-Bosch A, Cheng-Yang C, Tatti SA, Kasamatsu E, Iljazovic E, Odida M, Prado R, Seoud M, Grce M, Usubutun A, Jain A, Suarez GA, Lombardi LE, Banjo A, Menendez C, Domingo EJ, Velasco J, Nessa A, Chichareon SC, Qiao YL, Lerma E, Garland SM, Sasagawa T, Ferrera A, Hammouda D, Mariani L, Pelayo A, Steiner I, Oliva E, Meijer CJ, Al-Jassar WF, Cruz E, Wright TC, Puras A, Llave CL, Tzardi M, Agorastos T, Garcia-Barriola V, Clavel C, Ordi J, Andujar M, Castellsague X, Sanchez GI, Nowakowski AM, Bornstein J, Munoz N, Bosch FX; Retrospective International Survey and HPV Time Trends Study Group. Human papillomavirus genotype attribution in invasive cervical cancer: a retrospective cross-sectional worldwide study. Lancet Oncol. 2010 Nov;11(11):1048-56. doi: 10.1016/S1470-2045(10)70230-8. Epub 2010 Oct 15. PMID 20952254
- [Background] Franco EL, Villa LL, Sobrinho JP, Prado JM, Rousseau MC, Desy M, Rohan TE. Epidemiology of acquisition and clearance of cervical human papillomavirus infection in women from a high-risk area for cervical cancer. J Infect Dis. 1999 Nov;180(5):1415-23. doi: 10.1086/315086. PMID 10515798
- [Background] Munoz N, Mendez F, Posso H, Molano M, van den Brule AJ, Ronderos M, Meijer C, Munoz A; Instituto Nacional de Cancerologia HPV Study Group. Incidence, duration, and determinants of cervical human papillomavirus infection in a cohort of Colombian women with normal cytological results. J Infect Dis. 2004 Dec 15;190(12):2077-87. doi: 10.1086/425907. Epub 2004 Nov 22. PMID 15551205
- [Background] Shankar AH, Prasad AS. Zinc and immune function: the biological basis of altered resistance to infection. Am J Clin Nutr. 1998 Aug;68(2 Suppl):447S-463S. doi: 10.1093/ajcn/68.2.447S. PMID 9701160
- [Background] Al-Gurairi FT, Al-Waiz M, Sharquie KE. Oral zinc sulphate in the treatment of recalcitrant viral warts: randomized placebo-controlled clinical trial. Br J Dermatol. 2002 Mar;146(3):423-31. doi: 10.1046/j.1365-2133.2002.04617.x. PMID 11952542
- [Background] Simonart T, de Maertelaer V. Systemic treatments for cutaneous warts: a systematic review. J Dermatolog Treat. 2012 Feb;23(1):72-7. doi: 10.3109/09546634.2010.500324. Epub 2010 Nov 6. PMID 21054194
- [Background] Stefani M, Bottino G, Fontenelle E, Azulay DR. Efficacy comparison between cimetidine and zinc sulphate in the treatment of multiple and recalcitrant warts. An Bras Dermatol. 2009 Jan-Feb;84(1):23-9. doi: 10.1590/s0365-05962009000100003. English, Portuguese. PMID 19377755
- [Background] Kim JH, Bae SN, Lee CW, Song MJ, Lee SJ, Yoon JH, Lee KH, Hur SY, Park TC, Park JS. A pilot study to investigate the treatment of cervical human papillomavirus infection with zinc-citrate compound (CIZAR(R)). Gynecol Oncol. 2011 Aug;122(2):303-6. doi: 10.1016/j.ygyno.2011.04.026. Epub 2011 May 24. PMID 21605892
- [Background] Bulkmans NW, Berkhof J, Bulk S, Bleeker MC, van Kemenade FJ, Rozendaal L, Snijders PJ, Meijer CJ; POBASCAM Study Group. High-risk HPV type-specific clearance rates in cervical screening. Br J Cancer. 2007 May 7;96(9):1419-24. doi: 10.1038/sj.bjc.6603653. Epub 2007 Mar 6. PMID 17342094
- [Background] Nobbenhuis MA, Helmerhorst TJ, van den Brule AJ, Rozendaal L, Voorhorst FJ, Bezemer PD, Verheijen RH, Meijer CJ. Cytological regression and clearance of high-risk human papillomavirus in women with an abnormal cervical smear. Lancet. 2001 Nov 24;358(9295):1782-3. doi: 10.1016/S0140-6736(01)06809-X. PMID 11734239
- [Background] Lopez-Garcia DR, Gomez-Flores M, Arce-Mendoza AY, de la Fuente-Garcia A, Ocampo-Candiani J. Oral zinc sulfate for unresponsive cutaneous viral warts: too good to be true? A double-blind, randomized, placebo-controlled trial. Clin Exp Dermatol. 2009 Dec;34(8):e984-5. doi: 10.1111/j.1365-2230.2009.03623.x. No abstract available. PMID 20055878
- [Background] Fosmire GJ. Zinc toxicity. Am J Clin Nutr. 1990 Feb;51(2):225-7. doi: 10.1093/ajcn/51.2.225. PMID 2407097
- [Background] Molano M, Van den Brule A, Plummer M, Weiderpass E, Posso H, Arslan A, Meijer CJ, Munoz N, Franceschi S; HPV Study Group. Determinants of clearance of human papillomavirus infections in Colombian women with normal cytology: a population-based, 5-year follow-up study. Am J Epidemiol. 2003 Sep 1;158(5):486-94. doi: 10.1093/aje/kwg171. PMID 12936904
- [Background] Raza N, Khan DA. Zinc deficiency in patients with persistent viral warts. J Coll Physicians Surg Pak. 2010 Feb;20(2):83-6. PMID 20378032
- [Background] Miranda PM, Silva NN, Pitol BC, Silva ID, Lima-Filho JL, Carvalho RF, Stocco RC, Becak W, Lima AA. Persistence or clearance of human papillomavirus infections in women in Ouro Preto, Brazil. Biomed Res Int. 2013;2013:578276. doi: 10.1155/2013/578276. Epub 2013 Nov 5. PMID 24298551